CLINICAL TRIAL: NCT04836026
Title: Evaluation of the HF20™ Filter for Pediatric Continuous Renal Replacement Therapy (CRRT)
Brief Title: Registry for HF20 for Pediatric CRRT Under Emergency Use Authorization
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Stuart Goldstein, MD, Director, Center for Acute Care Nephrology, Children's Hospital Medical Center, Cincinnati
Other Study IDs: HF20 Registry
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Kidney Disease; Acute Kidney Injury
Keywords: HF20
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HF20™ for Pediatric CRRT: Pediatric patients in an intensive care unit requiring CRRT for acute kidney injury (AKI)
  Interventions: Device: HF20™

INTERVENTIONS:
Device: HF20™ — HF20™ will be used for CRRT

SUMMARY:
Historically, innovations for acute kidney injury (AKI) and continuous renal replacement therapy (CRRT) have centered around an adult population. However, research has shown that over 10% of pediatric patients develop severe AKI within the first week in an intensive care unit (ICU). When a pediatric patient requires renal replacement therapy for AKI in the ICU, CRRT is usually the modality of choice. The HF20™ is indicated for supporting patients weighing 8 to 20 kilograms, addressing a critical clinical need for critically ill children who require CRRT. Current US Food and Drug Administration (FDA) approved CRRT filters are designed for patients weighing more than 20 kg or less than 10 kg, leaving a gap in appropriately designed filters for pediatric patients.

A previous trial in the US showed that the HF20™ is safe and effective, however the membrane composition of the HF20™ used in that trial is different than what is currently manufacturer and available. Baxter Healthcare Corporation has received an Emergency Use Authorization (EUA) for the currently available HF20™ to be used in the era of the COVID-19 pandemic, however participants do not need to be infected with the SAR-CoV-2 virus in order to be treated. The EUA for the HF20™ allows for treatment for any children weighing between 8 and 20 kilograms in need of CRRT. This registry will collect clinical data related to the safety and efficacy of the HF20™ filter for CRRT in pediatric patients weighing 8 to 20 kilograms at participating institutions, however participation in this registry is not a requirement in order to be treated with the HF20™ filter.

ELIGIBILITY:
Inclusion Criteria:

* Receiving or plan to receive CRRT with the HF20™ filter as standard of care
* Acute kidney injury (AKI) or fluid overload as defined as one of the two below:

  1. AKI defined as Kidney Disease Improving Global Outcomes (KDIGO) Stage 1 or higher by either:

     1. Serum creatinine criteria (0.3 mg/dL increase over baseline in 48 hours, or a 50 percent increase within the previous 7 days) or
     2. Urine output criteria (less than 0.5 mL/kg/hr for 6 or more hours)
  2. Severe fluid overload defined as greater than 10 percent fluid accumulation based on ICU admission weight

Exclusion Criteria:

* Weight less than 8 kilograms
* Weight more than 20 kilograms
* Patient not expected to survive more than 48 hours
* Received renal replacement therapy in the previous 5 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving CRRT with the HF20™ filter as their standard care for AKI or fluid overload in an intensive care unit at a participating institution.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Blood Urea Nitrogen (BUN) | After 24 hours of CRRT with the HF20™ filter as compared to baseline

SECONDARY OUTCOMES:
Change in Serum Creatinine | After 24 hours of CRRT with the HF20™ filter as compared to baseline
Change in Serum Bicarbonate/Carbon Dioxide | After 24 hours of CRRT with the HF20™ filter as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No